CLINICAL TRIAL: NCT05868291
Title: Daylight-controlled Lighting Adjusted for Geographical Orientation : Effects on Recovery, Energy Consumption and User Satisfaction
Acronym: DIM Light
Status: Active, not recruiting | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Elforsk (Unknown)
Responsible Party: Sponsor
Other Study IDs: DIM Light
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Light
Keywords: DIM Light; Sleep; Energy Consumption; Chronotherapeutics; Built environment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: During the period going from November 2022 to March 2023, data from all the patients (approx. 500) hospitalized in the 4 closed wards will be collected (duration of stay, medication use...).
  The group 1 will be exposed to the standard lighting system in Bispebjerg Hospital.
- Group 2: During the period going from November 2023 to March 2024, data from all the patients (approx. 500) hospitalized in the 4 closed wards will be collected (duration of stay, medication use...).
  The group 2 will be exposed to the new lighting system that will have been optimized (higher intensity and blue content in the morning and progressively dimmed light after 14:00).

SUMMARY:
The trial takes place in 4 psychiatric closed wards at Ny Psykiatri Bispebjerg. The objective is to compare, retrospectively, over two consecutive winter periods (2022 and 2023) the effect of the lighting on the duration of stay of the patients. During the first winter, a standard lighting is used, and, during the second winter, the lighting will be modified to favor a greater light intensity in blue wave color light in the morning and a gradual decrease in light intensity in the evening adjusted for geographical orientation of the patients' rooms.

DETAILED DESCRIPTION:
Light has benefits in many pathologies, especially in psychiatry and sleep disorders. It is the most powerful Zeitgeber, allowing a drive of the sleep-wake rhythm. But what are the "doses or quantities" of light necessary for humans to stimulate circadian regulation? And how is it possible to promote better people's exposure to this amount of light during winter (especially in Nordic countries where daily light exposure during winter is particularly reduced: 8 hours on average)? At the Bispebjerg Hospital, following the installation of LED lighting, a dynamic system favoring a greater light intensity in blue wave color light in the morning and a gradual decrease in light intensity in the evening adjusted for geographical orientation of the patients' rooms is evaluated. This device was effective on anxious and depressive symptoms for patients hospitalized after a stroke. Here, we'll study the effect the light may have on patients in psychiatric closed wards. Moreover, we'll assess the users' satisfaction and the energy consumption of the system.

If the described intervention is associated with a reduction in the duration of stay of the patients in the ward as well as with a general satisfaction of the users and that it consumes much less energy, one could think of the installation of this system on a large scale not only in hospitals but also in schools or other public buildings where it could be interesting to have this adapted lighting.

ELIGIBILITY:
Inclusion Criteria:

* patients being 18 years old or older
* patients having a duration of stay of at least 3 days in the wards

Exclusion Criteria:

* patients that have switched room during their stay
* patients that have been in rooms where the lighting wasn't working

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above 18 years old that have been hospitalized in one of the 4 closed wards of NPB during the 2 study periods.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Duration of stay | The 2 periods consecutive winter period (2022 and 2023)
  Number of day of the stay of the partient in the closed ward of NPB (Ny Psykiatri Bispebjerg)

SECONDARY OUTCOMES:
Use of psychotropic medication | The 2 periods consecutive winter period (2022 and 2023)
  The mean use of psychotropic medication (in mg/day) during the two periods

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Ny Psykiatri Bispebjerg, Copenhagen, Region Sjælland
  - Mental Health Centre Copenhagen, Copenhagen

REFERENCES:
- [Derived] Volf C, Corell DD, Hansen TS, Dubois JM, Zeng X, Baandrup L, Petersen PM, Martiny K. Effects of dim-evening lighting optimised for geographical orientation versus standard lighting on mental health: protocol paper for a quasiexperimental study in a psychiatric hospital. BMJ Open. 2024 Oct 10;14(10):e086658. doi: 10.1136/bmjopen-2024-086658. PMID 39389598